CLINICAL TRIAL: NCT03742492
Title: Bioavailability of EPA + DHA Enriched Canned Tuna and Its Acute Effects on Cardiovascular Risk Markers, in Healthy Human Volunteers
Brief Title: Bioavailability of EPA + DHA Enriched Canned Tuna and Its Acute Effects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other); NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FUNCTIONALTUNA1
Record Dates: First submitted 2018-11-06; First posted 2018-11-15 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers
Keywords: Omega-3 fatty acids; Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA); Bioavailability; Blood pressure; Lipid absorption; Canned tuna
MeSH Terms: interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canned tuna + fish oil (5 g EPA + DHA) (Experimental): Meal containing canned tuna + fish oil (5 g EPA + DHA)
  Interventions: Dietary Supplement: Meal containing canned tuna + fish oil (5 g EPA + DHA)
- Canned tuna + soybean oil (Placebo Comparator): Meal containing canned tuna + soybean oil
  Interventions: Dietary Supplement: Meal containing canned tuna + soybean oil

INTERVENTIONS:
Dietary Supplement: Meal containing canned tuna + fish oil (5 g EPA + DHA) — Meal containing canned tuna + fish oil (5 g EPA + DHA)
  Arms: Canned tuna + fish oil (5 g EPA + DHA)
Dietary Supplement: Meal containing canned tuna + soybean oil — Meal containing canned tuna + soybean oil
  Arms: Canned tuna + soybean oil

SUMMARY:
Evidence has suggested that omega-3 fatty acids, namely eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), have an important role in promoting cardiovascular health. However, the currently available scientific literature describing the postprandial effects and bioavailability of these fatty acids, particularly when they are incorporated into high protein food item, like canned tuna, is far from conclusive.

The aim of this study is to evaluate the acute bioavailability of EPA + DHA enriched canned tuna and its acute effects on cardiovascular risk markers, in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women
* Age 18 - 59 years
* Willing to maintain usual diet and physical activity patterns
* Willing to comply with study protocol and procedures
* Willing to provide written informed consent

Exclusion Criteria:

* Pregnant, breastfeeding or planning to become pregnant within the study period
* Subjects with current or previous cardiovascular disease (ischemic cardiovascular disease, angina stable or unstable; myocardial infarction, stroke or symptomatic peripheral arteriosclerosis)
* Subjects with liver or kidney diseases or cancer
* Diabetes mellitus (fasting glycemia> 126 mg / dL)
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg)
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to cooperate during the study
* Subjetcs with gastrointestinal disorder or under prescription for medication affecting gastrointestinal function or absorption of nutrients
* Known allergy (or sensitivity) to omega-3 fatty acids, fish (tuna), crustaceans, lactose or any meal ingredient
* With antihypertensive therapy
* Health condition that prevents compliance with study requirements
* Subjects under prescription for medication for digestive symptoms such as anti-spasmodic, laxatives and anti-diarrheic drugs or other digestive auxiliaries
* Subjects under prescription of anticoagulant drugs
* Dietary patterns or supplement use that could interfere with study evaluations
* Subjects not willing to avoid the consumption of fish oil or food supplements, including fatty acids, during the study (except as indicated in the study protocol)
* Use of antibiotics in the last 4 weeks and laxatives in the last 2 weeks

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial plasma triglycerides concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of triglycerides (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma low-density lipoprotein (LDL) cholesterol concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of LDL cholesterol (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma total cholesterol concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of total cholesterol (0, 1, 2, 3, 4, and 5 hours post-meal).

SECONDARY OUTCOMES:
Change in postprandial blood pressure | Up to 5 hours post-meal.
  Impact on the postprandial levels of blood pressure (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma high-density lipoprotein (HDL) cholesterol concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of HDL cholesterol (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma eicosapentaenoic acid (EPA) concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of EPA (0, 2, 4, and 5 hours post-meal).
Change in postprandial plasma docosahexaenoic acid (DHA) concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of DHA (0, 2, 4, and 5 hours post-meal).
Change in postprandial plasma blood glucose concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of blood glucose (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma insulin concentrations | Up to 5 hour post-meal.
  Impact on the postprandial levels of insulin (0, 1, 2, 3, 4, and 5 hours post-meal).
Change in postprandial plasma Apolipoprotein B-48 (apoB-48) concentrations | Up to 5 hours post-meal.
  Impact on the postprandial levels of ApoB-48 (0, 1, 2, 3, 4, and 5 hours post-meal).

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS, NOVA Medical School; Luís Azevedo, PhD, Principal Investigator — CINTESIS, Faculty of Medicine of the University of Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project FUNCTIONALTUNA financed by COMPETE2020 (POCI-01-0247-FEDER-003466) — https://www.researchgate.net/project/FUNCTIONALTUNA